CLINICAL TRIAL: NCT00568854
Title: Converging Epidemics: Immunobiology of Diabetes Mellitus and Tuberculosis Infection
Brief Title: Immunobiology of Diabetes and Tuberculosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Additional funding was not secured
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alicia H. Chang, MD, Instructor, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SU-10182007-744
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-06

CONDITIONS: Tuberculosis; Diabetes Mellitus
MeSH Terms: conditions — Tuberculosis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Participants with diabetes (Active Comparator): Persons with diagnosis of diabetes. Received biological intervention: BCG
  Interventions: Biological: BCG
- Participants without diabetes (Active Comparator): Persons with no diagnosis of diabetes and negative diabetes screening labs. Received biological intervention: BCG.
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: BCG — Both arms: diabetics and nondiabetics will receive vaccination in the upper arm with a 0.1-mg intradermal dose of a single strain of BCG (Mycobax, Sanofi-Aventis), which is FDA approved for this indication.

SUMMARY:
The study hypothesis is that type 2 diabetics have abnormal cell-mediated immunity to tuberculosis manifesting as altered cytokine responses by peripheral blood mononuclear cells (PBMCs). This hypothesis will be tested using the live tuberculosis vaccine, Bacille Calmette-Guerin (BCG), in U.S.-born type 2 diabetics and nondiabetics. The investigators will control for potential confounding by age, sex, race, comorbidities, and select medications. Expression of key cytokines will be measured with real-time polymerase chain reaction.

DETAILED DESCRIPTION:
The project has three specific aims:

Specific Aim 1: To assess differences between the study groups in cytokine expression before and after BCG vaccination. The investigators will determine within-individual variability in cytokine measurements and describe the kinetics of cytokine response to BCG. Peak response levels, time to peak, and patterns of cytokines expressed will be compared.

Specific Aim 2: To evaluate the effect of hyperglycemia on the cytokine response of type 2 diabetics. The investigators will evaluate whether levels of hemoglobin A1C (HbA1C) are associated with degree of cytokine response and test if type 2 diabetics who have good glucose control are different from nondiabetics.

Specific Aim 3: To evaluate the effect of testing PBMCs from diabetics outside of their diabetic milieu. Investigators will compare the BCG-specific cytokine responses of PBMCs stimulated in normal medium, PBMCs stimulated in glucose correlating to the person's most recent HbA1C, and whole blood samples.

ELIGIBILITY:
Inclusion Criteria:Type 2 diabetes or healthy individual Able to give consent US-born Age 30-65 Exclusion Criteria:* Immunosuppressive disease

* Immunosuppressive medications
* Pregnancy
* Renal failure
* Advanced pulmonary disease
* Prior BCG vaccination
* Prior TB infection
* Type 1 diabetes

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Hsin-Ming Chang, Sub-Investigator — Stanford University; Julie Parsonnet, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Diabetes | Participants Without Diabetes
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Diabetes | Participants Without Diabetes | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Median (Full Range); unit: years] | 59.5 [54 to 65] | 41.5 [32 to 46] | 54.5 [32 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Hemoglobin A1C [Median (Full Range); unit: %] | 6.65 [6.1 to 7.5] | 5.65 [5.6 to 5.7] | 6.1 [5.6 to 7.5]

OUTCOME MEASURES:

1. Primary Outcome: Antigen-specific Immune Response Measured by Reaction to Tuberculin Skin Test
Description: Participants had baseline tuberculin testing (TST), followed by BCG vaccination, and at 5 months after vaccination, study participants had repeat tuberculin skin testing done.
Time Frame: 5 months
Measure: Median (Full Range); unit: mm
Arm/Group | Participants With Diabetes | Participants Without Diabetes
Number analyzed (Participants) | 6 | 4
mm | 0 [0 to 10] | 3 [0 to 6]

2. Primary Outcome: Kinetics of Mycobacterial-specific Immune Response After BCG Vaccination
Description: Blood was sampled at times 0, 2, 4, 6, 8, 12, 16, and 20 weeks post BCG vaccination and Interferon gamma production was measured as change from pre-vaccination baseline. Timeline of peak IFn-g response was measured for both study groups.
Time Frame: 5 months
Measure: Mean (Standard Deviation); unit: weeks when peak response was observed
Arm/Group | Participants With Diabetes | Participants Without Diabetes
Number analyzed (Participants) | 6 | 4
weeks when peak response was observed | 8 (1) | 8 (1)

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Participants With Diabetes | Participants Without Diabetes
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

LIMITATIONS AND CAVEATS:
This was a pilot/feasibility study to lay groundwork for a larger scale study of differences in immune responses in persons with diabetes versus persons without diabetes. The study aimed to optimize laboratory procedures for the full study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No